CLINICAL TRIAL: NCT01916122
Title: Fluorestradiol (FES) PET/CT for Imaging Estrogen Receptor Status
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-071
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Fluorestradiol (FES); PET/CT scan; Estrogen Receptor; 13-071
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- (FES) PET/CT for Imaging (Experimental): FES PET/CT studies will be performed as hybrid PET/CT examinations for attenuation correction and lesion localization. A bolus of 5 mCi (+/- 10%) of FES PET/CT will be injected intravenously. 60 (+/- 10) minutes following tracer injection, the patient will be positioned on a GE Discovery PET/CT scanner. A low milliampere CT of from the mid skull to mid thigh will be acquired first, 60-80mAs, 120-140kVp, with a 5mm slice thickness while the patient was free breathing. PET will be acquired at 3-5 minutes per bed position using the 3D mode, approximately 6-7 bed positions. FES PET/CT imaging will take less than 60 minutes. Scans will be reconstructed with iterative reconstruction.
  If follow-up FES PT/CT scans are performed on a patient, then the same parameters will be used as the initial FES PET/CT scan.
  Interventions: Drug: Fluorestradiol (FES); Procedure: PET/CT Imaging

INTERVENTIONS:
Drug: Fluorestradiol (FES)
Procedure: PET/CT Imaging

SUMMARY:
These are tumors which expresses estrogen receptors. Estrogen receptors are found within breast cancer cells and are an important marker of which medicines may best treat a breast cancer. This study is being performed to imaging the amount of estrogen receptors expressed in the tumor. A research agent named 16α-18F-fluoroestradiol (FES) finds estrogen receptors and binds to them. Then tumors with estrogen receptors can be imaged by a PET/CT scanner, a machine that can take pictures of where the FES is and how much FES is present. The results of this study may help researchers know whether FES can be used to monitor changes in estrogen receptors in tumors during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic/immunochemical proof of ER+ primary or metastatic malignancy (positive staining in ≥ 1% of cells by immunohistochemistry).
* Patients who are to be treated with clinically approved or experimental regimens where ER has an important role
* ECOG performance status of 0-2.
* Patients must provide written informed consent

Exclusion Criteria:

* Age <18 years
* Patients who cannot undergo PET/CT scanning (i.e. because of weight limits, claustrophobia)
* Pregnancy or lactation
* Total serum bilirubin > 1.5 times upper limit of normal (abnormal hepatic metabolism may interfere with FES hepatic excretion). Increased serum bilirubin due to Gilbert's syndrome is permitted.
* Serum creatinine > 1.5 times upper limit of normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
FES PET/CT scanning | 5 years
  The objective of this study is only to allow FES PET/CT scanning of patients at MSKCC. This protocol is an "umbrella protocol" to allow FES PET/CT scanning to be used in other companion protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Randy Yeh, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/